CLINICAL TRIAL: NCT06094309
Title: Randomized Pilot Study Evaluating Effectiveness of Botulinum Toxin Type A in Freezing Walking in Parkinson's Disease
Brief Title: Effectiveness of Botulinum Toxin in Freezing of Gate in Parkinson's Disease Walking in Parkinson's Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centro Hospitalar de Lisboa Central (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHULC.CI.431.2022
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Freezing of Gate; Parkinson Disease; Botulinum Toxin
MeSH Terms: conditions — Parkinson Disease | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: botulinum toxin (Active Comparator): The botulinum toxin injection will be carried out by a doctor with experience in this therapeutic modality, which in turn is not part of the group of doctors who observe patients in the initial and subsequent phases. 100 Units (U) of botulinum toxin type A, in each lower limb (200 U in total), in muscle proximal thigh, once, at a moment that will be defined as T0. This group of 10 participans.
  Interventions: Drug: Botulinum toxin type A injection
- Active Comparator: Placebo (Placebo Comparator): In the control group, patients will be subject to the same protocol, with the difference in that the injections will be saline, although they look the same on the outside. You doctors carrying out therapy and evaluating progress during face-to-face visits will not have access to the distribution of groups. This group of 10 participans.
  Interventions: Drug: Botulinum toxin type A injection

INTERVENTIONS:
Drug: Botulinum toxin type A injection — The BT injection will be performed by a doctor with experience in this therapy, with 100 Units (U) of type A BT, bilaterally, in the flexor muscle of the thigh, once, with replacement of the same ampoules with saline in controls. To the Patient assessments will take place over 4 months, weekly by telephone using a questionnaires on freezing and the notion of clinical improvement (FOGQ and SCGIC, respectively) and monthly in person with objective assessments using the MDS-UPDRS scales - part III motor assessment, Timed Up & Go and Two Minute Walk.

SUMMARY:
Freezing of gait is a symptom of Parkinson's disease (PD) that becomes more evident with the evolution of the disease, and which presents an important difference compared to the other signs and symptoms: does not respond adequately to dopaminergic therapy, which calls into question its pathophysiology. In this sense, and through empirical experience, it has been noted that freezing responds to cueing techniques (visual, sensory motor, auditory tricks, among others) which suggests a similarity with dystonic pathology. This similarity could be the basis of a common response to botulinum toxin (BT). Objectives: This study aims to understand whether BT is an effective therapy for freezing gait in patients with Parkinson's disease. Methodology: This is a prospective parallel study with therapeutic intervention, controlled by placebo, double blind. The randomization of groups will be stratified. The population will be recruited from from the CHLC movement disorders consultation, and that meets the following inclusion criteria: Parkinson's disease with freezing of gait, scoring > 1 at point 2.13 on the scale MDS-UPDRS and be responsive to cueing techniques, with severity of Parkinson's disease rated 3 or 4 on the Hoehn & Yahr scale. The BT injection will be performed by a doctor with experience in this therapy, with 100 Units (U) of type A BT, bilaterally, in the flexor muscle of the thigh, once, with replacement of the same ampoules with saline in controls. To the Patient assessments will take place over 4 months, weekly by telephone using a questionnaires on freezing and the notion of clinical improvement (FOGQ and SCGIC, respectively) and monthly in person with objective assessments using the MDS-UPDRS scales - part III motor assessment, Timed Up & Go and Two Minute Walk.

DETAILED DESCRIPTION:
Study with therapeutic intervention, placebo-controlled, double-blind, with stratified randomization using the minimization method. The variables to consider by this method will be binary variables and three will be considered: the severity of the freezing (degree 2 freezing / degree 3 and 4 freezing)8, the severity of the disease Parkinson's (Hoehn & Yahr (H&Y) stage 3 / H&Y stage 4)9 and cognitive capacity (Mini-Mental State Examination (MMSE) 10-23 / MMSE 24-30)10.

People with Parkinson's disease in advanced stages, with freezing of gait frequent, responsive to cueing techniques, followed in consultation for diseases of the movement at CHULC, with the participation of doctors specializing in diseases of movement. All eligible participants will be required to complete the consent informed prior to their inclusion in the study.

Inclusion criteria: people with idiopathic Parkinson's disease with the presence of gait freezing, which scores > 1 at point 2.13 of the MDS-UPDRS8 scale and is responsive to cueing techniques, with severity of Parkinson's disease classified between 3 and 4 on the Hoehn & Yahr9 scale.

Exclusion criteria: previous exposure to toxin therapy, alteration of therapy for PD during the course of the study, cognitive impairment with MMSE10 < 10.

There will be two distinct modalities of observation and assessment of patients: in person, every month for 4 months, with observation of the patient and application of MDS-UPDRS8 scale, Timed Up & Go (TUG) scale11, and Two Minutes Walk scale12 and telephone, every week for 4 months, with the application of a questionnaire on the freezing and another about the impression of improvement. Both assessment modalities will be carried out by doctors from the Neurology service.

1. Observation of the patient before administration of BT therapy and every month, on a scheduled basis, at the same time, 12 hours after suspension of the levodopa therapy (T0, T1M, T2M, T3M, T4M) and classification of scales Timed Up & Go11 and Two Minutes Walk12;
2. Application of the FOGQ13 and SCGIC14 questionnaires before administration of the therapy and every week, via telephone, to the patient (T0, T1S, T2S, T3S, T1M, T5S, T6S, T7S, T2M, T9S, T10S, T11S, T3M, T13S, T14S, T15S, T4M).

ELIGIBILITY:
Inclusion Criteria: people with idiopathic Parkinson's disease with the presence of gait freezing, which scores > 1 at point 2.13 of the MDS-UPDRS8 scale and is responsive to cueing techniques, with severity of Parkinson's disease classified between 3 and 4 on the Hoehn & Yahr9 scale.

Exclusion Criteria: previous exposure to toxin therapy, alteration of therapy for PD during the course of the study, cognitive impairment with MMSE10 < 10.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Variation Unified Parkinson's Disease Rating Scale (MDS-UPDRS8) | for 4 months after the study
  which is defined as fever (auricular temperature >38ºC) and elevation of CRP (> 75 mg/L), during the first 3 days after operation.
Variation Escala "Timed Up & Go"11 | for 4 months after the study
  20% improvement in completion time in any reevaluations;
Variation Escala Two Minutes Walk12 | for 4 months after the study
  20% improvement in the distance covered in any reevaluations;

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Margarida Grilo da Silva Dias, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No